CLINICAL TRIAL: NCT06331767
Title: mSYNC: an mHealth SYNdemic-based Consultation-liaison HIV Prevention Intervention for the Emergency Department
Brief Title: Development of a Multilevel HIV Prevention Intervention for the Emergency Department
Acronym: mSYNC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Tiffany R. Glynn, PhD, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024P000654; K23DA060719 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-03-26 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: HIV; Drug Use; Mental Health; Psychological Distress; Social Marginalization; Problems With Access to Health Care
MeSH Terms: conditions — Psychological Well-Being; Social Marginalization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- mSYNC (Experimental): mHealth psychosocial-behavioral intervention
  Interventions: Behavioral: mSYNC

INTERVENTIONS:
Behavioral: mSYNC — mSYNC in an mHealth HIV prevention intervention to be initially delivered at point-of-care during a visit to the emergency department with continued on demand access to intervention app at home. Taking a behavioral medicine approach, mSYNC simulates hospital-based consultation & liaison psychology service by intervening on interrelated health risk behaviors, mental health issues, and structural/treatment needs. The mHealth app includes modules with motivational interviewing for HIV/drug use risk behaviors, cognitive behavioral therapy for transdiagnostic psychological coping skills, referral system for needed hospital-based services (mental health/drug use treatment; HIV prevention; social services), and access to geolocated resources.

SUMMARY:
The goal of this clinical trial is to pilot test a psychosocial-behavioral mobile health (mHealth) human immunodeficiency virus (HIV) prevention intervention in people who use drugs presenting to the emergency department (ED). The main question the study aims to answer is: is the intervention acceptable and appropriate? Participants will use the mHealth app while waiting in the ED and also at home for 90 days. Participants will be asked to complete surveys at baseline, before leaving the ED, and at 30-, 60-, and 90-day follow up visits.

DETAILED DESCRIPTION:
"mSYNC" (mHealth SYNdemic-based Consultation & liaison) is an mHealth HIV prevention intervention to be initially delivered at point-of-care during a visit to the emergency department with continued on demand access to intervention app at home. mSYNC simulates hospital-based consultation and liaison psychology service by intervening on the interrelated health risk behaviors, mental health issues, and structural/treatment needs (e.g., housing, drug use treatment). Capitalizing on the syndemic domino effect, mSYNC aims to promote prevention via entry into at least one of three interacting pathways: decreased HIV/drug use risk behaviors, decreased severity of mental health symptoms, and increased linkage to services. A pilot single-arm feasibility test will be conducted to assess patient-level implementation outcomes of acceptability and appropriateness of the mHealth intervention. Secondarily, change over time will be explored for HIV risk, drug use, mental health symptoms, and linkage to care. The study will take place in two urban emergency departments in Boston, Massachusetts. A sample of N=100 people who use drugs (PWUD) who also belong to other key HIV risk groups (transgender women, men who have sex with men [MSM], Black/Latinx/Indigenous people) will be enrolled during a visit to the emergency department. Research staff will pre-screen individuals checked-in and waiting in the emergency department for potential eligibility via information from electronic medical chart (HIV risk or drug use indicator). Staff will then approach potentially eligible patients identified from this pre-screen to describe the study and invite them to be screened for eligibility. Once screened eligible, participants will complete a baseline survey and asked to engage with the mHealth intervention app during their time in the ED (environment- and person-driven intervention dosage). Before discharge, participants will complete a brief feedback survey and asked to use to mHealth at home for at least one time a week for the next 90 days (environment- and person-driven intervention dosage) with the help of automatic notifications personalized to the person. Participants will complete a remote follow-up at 30, 60, and 90 days consisting of a quantitative survey and exit interview (90-day follow-up only).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* No HIV positive test in electronic medical record or self-reported
* Past month HIV risk behavior (condomless sex or needle sharing not protected by adherent PrEP [pre-exposure prophylaxis])
* Past month use of illicit drugs (excluding marijuana)
* Belong to at least one of key HIV risk group (transgender woman, MSM, Black/Latinx/Indigenous)
* Own a smartphone
* Able to read and understand English

Exclusion Criteria:

* Unable to provide informed consent
* Medical or psychiatric condition that would interfere with ability to participate in study procedures
* Presented to the emergency department (ED) for a psychiatric issue
* Expected to be admitted to ED for more than 48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Acceptability of intervention assessed via AIM | immediate post intervention exposure, 90-day follow-up
  The Acceptability of Intervention Measure (AIM) is a 4-item Likert agreeability scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated resulting in a continuous score with higher scores indicating greater intervention acceptability.
Acceptability: Usability of mHealth intervention assessed via SUS | immediate post intervention exposure, 90-day follow-up
  The System Usability Scale (SUS) is a 10-item Likert agreeability scale ranging from 1 (Strongly disagree) to 5 (Strongly agree). Scoring results in a continuous score ranging from 0 to 100 with higher scores indicating greater intervention acceptability.
Acceptability of intervention assessed qualitatively | 90-day follow-up
  Qualitative exit interview will be structured on Proctor's implementation outcome definition for intervention acceptability (satisfaction with intervention content, complexity, comfort, delivery, and credibility)
Appropriateness of intervention assessed via IAM | immediate post intervention exposure, 90-day follow-up
  The Intervention Appropriateness Measure (IAM) is a 4-item Likert agreeability scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated resulting in a continuous score with higher scores indicating greater intervention appropriateness.
Appropriateness: Intervention engagement assessed via UES | immediate post intervention exposure, 90-day follow-up
  The User Engagement Scale (UES) is a 31-item Likert agreeability scale ranging from 1 (Completely disagree) to 5 (Completely agree). A mean score is calculated resulting in a continuous score with higher scores indicating greater intervention appropriateness.
Appropriateness of intervention assessed qualitatively | immediate post intervention exposure, 90-day follow-up
  Qualitative exit interview will be structured on Proctor's implementation outcome definition for intervention appropriateness (perceived fit of intervention: relevance, compatibility, suitability, usefulness, practicability).